CLINICAL TRIAL: NCT02122627
Title: Prevention of Exacerbations in Patients With COPD Through Vitamin D Supplementation: a Randomized Controlled Trial
Brief Title: Vitamin D Supplementation in Patients With COPD
Acronym: PRECOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Leiden University Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Renate T de Jongh, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5.1.13.033
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Vitamin D, COPD, immunomodulation, pulmonary function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): colecalciferol 16.800 IU per week
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — Colecalciferol 16.800 IU per week
  Other Names: Colecalciferol, cholecalciferol, vitamin D3
  Arms: Vitamin D
Drug: Placebo
  Arms: Placebo

SUMMARY:
Vitamin D has an immunomodulatory role. the aim of the present study is to assess the effect of vitamin D supplementation on exacerbation rate of COPD patient with a vitamin D deficiency.

DETAILED DESCRIPTION:
Rationale: Although vitamin D is well known for its function in calcium homeostasis and bone mineralisation, several studies have shown immunomodulatory effects of vitamin D. Vitamin D deficiency is a common problem in patients with COPD..

Objective: To assess the effect of vitamin D supplementation on exacerbation rate in patients with COPD and a vitamin D deficiency.

Study design: Randomized, multi-center, double-blind, placebo-controlled intervention study.

Study population: 240 patients aged 40 years and older with COPD and a vitamin D deficiency (25-hydroxyvitamin D concentration(25OHD)<50 nmol/l) with a COPD exacerbation. An exacerbation is defined as sustained worsening of respiratory symptoms during 48 hours and requiring oral corticosteroid, antibiotic or combination treatment that was initiated by a physician. Respiratory symptoms include at least one of the Anthonisen criteria (increased dyspnoea, sputum volume or purulence). Patients with a severe vitamin D deficiency (25OHD<15 nmol/l), known osteoporosis and/or use of vitamin D supplementation > 400 IU per day will be excluded.

Intervention: Participants will be randomly allocated to receive vitamin D3 16800 IU or placebo orally once a week during 1 year.

Main study parameters/endpoints: The primary endpoint is exacerbation rate.

Follow-up of the study:

Recruitment of participants is more troublesome than expected due to several reasons, more use of vitamin D supplements, higher 250hydroxyvitamin D levels than anticipated, less suitability due to presence other exclusion criteria.

29/8/2017 total number recruited participants is 119

10/7/2018 closure of recruitment, total number recruited participants is 158

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* aged above 40 years
* GOLD stages II-IV and diagnosis COPD confirmed by a medical doctor.
* minimum of 10 packyears of smoking
* vitamin D deficiency (a serum 25-hydroxyvitamin D lower than 50 nmol/l)
* ability to comply with all study requirements

Exclusion Criteria:

* pregnant or lactating women, or subjects who intend to become pregnant within the study period
* self-reported history of hypercalciemia or nephrolithiasis
* self-reported presence of sarcoidosis
* severe vitamin D deficiency (serum 25-hydroxyvitamin D lower than 15 nmol/l)
* life expectation of less than 6 months on the basis of concurrent disease
* interfering malignant diseases.
* diagnosed osteoporosis
* diagnosed asthma
* diagnosed chronic kidney disease stage 4 or higher (estimated glomerular filtration rate ≤ 29 ml/min/1,73 m2)
* serious mental impairment i.e. preventing to understand the study protocol or comply with the study aim; potentially unreliable patients and those judged by the investigator to be unsuitable for the study
* use of maintenance dose oral corticosteroids
* use of multivitamin supplement or vitamin D supplement which contains more than 400 IU per day
* current participation in a clinical rehabilitation programme

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Exacerbation rate | 1 year
  Definition of an exacerbation is according to the Anthonisen criteria

SECONDARY OUTCOMES:
Time to first and second exacerbation | 1 year
  Time to first and second exacerbation
Time to first hospitalisation | 1 year
  Time to first hospitalisation
FEV1 | 1 year
  Forced Expiratory Volume in 1 sec
IC | 1 year
  Inspiratory capacity
FEV1/FVC | 1 year
  Forced expiratory volume in 1 sec/ forced vital capacity
FRC | 1 year
  Functional residual capacity
RV | 1 year
  Residual volume
TLC | 1 year
  Total lung capacity
MIP | 1 year
  Maximal inspiratory pressure
MEP | 1 year
  Maximal expiratory pressure
SMWT | 1 year
  Six-minute walk test
Chair stand test | 1 year
  Chair stand test
3-meter walking test | 1 year
  3-meter walking test
Tandem stand test | 1 year
  Tandem stand test
Total score physical function tests | 1 year
  The sum score of the physical function tests
Hand grip strength | 1 year
  Hand grip strength
Quality of life (SGRQ) | 1 year
  QoL by the St George respiratory questionnaire
Quality of life (SF12) | 1 year
  QoL by the 12 item short form survey
Anxiety (HADS) | 1 year
  Anxiety by the hospital anxiety and depression scale
Depression (CESD) | 1 year
  Depression by the center for epidemiologic studies depression scale
Quality of life (CCQ) | 1 year
  QoL by the Clinical COPD Questionnaire score
Concentrations of antimicrobial peptides and pro-inflammatory mediators in nasal secretions | 1 year
  AMPs in nasal secretions
Ex-vivo cytokine production capacity of peripheral blood mononuclear cells and immunophenotyping | 1 year
  cytokine production capacity by PBMCs
Typing of bacteria and viruses in nasal secretions | 1 year
  Typing of bacteria and viruses in nasal secretions
Use of corticosteroids | 1 year
  Use of corticosteroids
Use of antibiotics | 1 year
  Use of antibiotics
Physical activity (SQUASH) | 1 year
  physical activity by short questionnaire to assess health-enhancing physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Martin den Heijer, Prof, Principal Investigator — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Radboud University Medical Center, Nijmegen

REFERENCES:
- [Background] Rafiq R, Aleva FE, Schrumpf JA, Heijdra YF, Taube C, Daniels JM, Lips P, Bet PM, Hiemstra PS, van der Ven AJ, den Heijer M, de Jongh RT. Prevention of exacerbations in patients with COPD and vitamin D deficiency through vitamin D supplementation (PRECOVID): a study protocol. BMC Pulm Med. 2015 Sep 23;15:106. doi: 10.1186/s12890-015-0101-4. PMID 26399451
- [Derived] Rafiq R, Aleva FE, Schrumpf JA, Daniels JM, Bet PM, Boersma WG, Bresser P, Spanbroek M, Lips P, van den Broek TJ, Keijser BJF, van der Ven AJAM, Hiemstra PS, den Heijer M, de Jongh RT; PRECOVID-study group. Vitamin D supplementation in chronic obstructive pulmonary disease patients with low serum vitamin D: a randomized controlled trial. Am J Clin Nutr. 2022 Aug 4;116(2):491-499. doi: 10.1093/ajcn/nqac083. PMID 35383823